CLINICAL TRIAL: NCT03977506
Title: Study of the Metrological Properties of Two Assessment Grids of the Driving Capacity After a Cerebrovascular Accident :Recommendations of the HAS (Hight Autority of Health in France) and Test Ride for Investigation Practical Fitness to Drive
Brief Title: Study of the Metrological Properties of Two Assessment Grids of the Driving Capacity After a Cerebrovascular Accident (ROADTRIP)
Acronym: ROADTRIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of recrutment
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2016 BARDOUX; 2017-A02276-47 (Other: ANSM)
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: driving capacity; cerebrovascular accident; grid
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All the inclusive patients will benefit the first test of driving during 45minutes. The evaluation will be realized by a present occupational therapist and a neuropsychologist in the vehicle.
  The second test on road will be for the part of included patients and will be made with the driving instructor and the therapist.
  Then, the third test on road will be realized after sessions on driving simulator for the part of the patients requiring a re-entrainment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavoiral (Experimental): The evaluation will be realized on two different assessment grids during the test on the road
  Interventions: Diagnostic Test: On-road driving evaluation

INTERVENTIONS:
Diagnostic Test: On-road driving evaluation — The data assessed during the road test from the two assessment grids (recommendations of the HAS and Test ride for investigation practical fitness to drive) :
  road position, vehicle control, track management, safety distances, speed, visual behavior, traffic signs, vehicle overtaking, anticipatory reactions and capabilities adaptation, attentional skills, decision-making, communication with other road users, assessment of specific situations such as insertion on a 2x2 lane, mechanical management and general impressions.

SUMMARY:
Precise recommendations concerning the methods of evaluation for the resumption of the driving after a not evolutionary stroke were recommended recently by the High Authority of Health. These describe among others elements to be estimated during the test on the road, in the presence of the driving instructor who remains Gold standard.

However, no standardized assessment grid serving as decision-making tool is at present validated.

Actually the test made by the unit of evaluation of the automobile resumption of the university hospital on the road, in a car of apprenticeship with double pedals and in the presence of a professional binomial (driving instructor and occupational therapist) then validated by the opinion of the doctor of the service. The current standard is thus very subjective and lack of sensibility.

It is necessary to study the metrological properties of both available assessment grids (that established from the recommendations of the HAS and TRIP), none of them reached a level of validation enough in this population.

The TRIP is this day validated only at the elderly people. The hypothesis of the search is an insufficiency of TRIP to estimate the patients presenting aftereffects of cerebrovascular accident.

The main objective of this work is to validate the new assessment grid after a study of its metrological properties in the situation of the driving on the road.

DETAILED DESCRIPTION:
The patients will benefit a medical consultation to estimate the possibility of inclusion in the study. During this consultation, the results of the neuropsychological and ophthalmological examinations will be explored and a specificity of the sensitive-driving deficits presented by the patient will be estimated to recommend the arrangements of necessary vehicle if necessary.

All the inclusive patients will benefit then the first test of driving in "ecological" situation accompanied by a lasting driving instructor during 45minutes. The evaluation will be realized by a present occupational therapist and a neuropsychologist in the vehicle, on two different assessment grids.

The second test on road will be for the part of included patients and will be made with the driving instructor and the therapist.

Then, the third test on road will be realized after sessions on driving simulator for the part of the patients requiring a re-entrainment.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 80 Years
* Cognitive and/or sensitive-motor disorders after a cerebrovascular accident
* Candidate for resumption of driving on the road and having to pass an aptitude test
* French legal protection

Exclusion Criteria:

* Contraindications for resumption of driving on the road (visual field amputation, binocular visual acuity less than 5/10; cognitive impairment not compatible with driving; other medical contraindication).
* Protected populations not concerned by the study (guardianship, curatorship, deprived of the freedoms, safeguarding of justice).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
The metrologic properties of the two evaluation grids (evaluation grids based on HAS and TRIP recommendations) | at day 1
  Acceptability will be based on the calculation of missing data at the level of each item and for the overall score of the study grids. Internal Consistency will be determined through Cronbach's alpha coefficient. Internal validity will be determined by study of correlation between the domains composing of the HAS and TRIP grids. Reproducibility .the Kappa concordance correlation coefficient will be used to determine the test-retest reliability. Internal validity will be determined by study of the correlation between of HAS and TRIP grids. External validity will be based on the study of correlations of scores from HAS and TRIP grids (Pearson or Spearman according to statistical distribution).
The metrologic properties of the two evaluation grids (evaluation grids based on HAS and TRIP recommendations) | at 1 month
  Acceptability will be based on the calculation of missing data at the level of each item and for the overall score of the study grids. Internal Consistency will be determined through Cronbach's alpha coefficient. Internal validity will be determined by study of correlation between the domains composing of the HAS and TRIP grids. Reproducibility .the Kappa concordance correlation coefficient will be used to determine the test-retest reliability. Internal validity will be determined by study of the correlation between of HAS and TRIP grids. External validity will be based on the study of correlations of scores from HAS and TRIP grids (Pearson or Spearman according to statistical distribution).
The metrologic properties of the two evaluation grids (evaluation grids based on HAS and TRIP recommendations) | at 3 months
  Acceptability will be based on the calculation of missing data at the level of each item and for the overall score of the study grids. Internal Consistency will be determined through Cronbach's alpha coefficient. Internal validity will be determined by study of correlation between the domains composing of the HAS and TRIP grids. Reproducibility .the Kappa concordance correlation coefficient will be used to determine the test-retest reliability. Internal validity will be determined by study of the correlation between of HAS and TRIP grids. External validity will be based on the study of correlations of scores from HAS and TRIP grids (Pearson or Spearman according to statistical distribution).

SECONDARY OUTCOMES:
The sensitivity to change | at 3 months
  The ability of the instrument to highlight a variation deemed relevant by experts, will be explored. The analyses described above for the tests-retest comparisons analyses will be re-implemented, the calculation of the effect-size will be performed for each grid
The sensitivity to change | at day 1
  The ability of the instrument to highlight a variation deemed relevant by experts, will be explored. The analyses described above for the tests-retest comparisons analyses will be re-implemented, the calculation of the effect-size will be performed for each grid
The sensitivity to change | at 1 month
  The ability of the instrument to highlight a variation deemed relevant by experts, will be explored. The analyses described above for the tests-retest comparisons analyses will be re-implemented, the calculation of the effect-size will be performed for each grid

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bardoux, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France